CLINICAL TRIAL: NCT02408588
Title: Evaluation of Compensatory Reserve in Obstetrical Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1996
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Parturition; Fetal Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Childbirth and epidural: Pregnant women giving childbirth who receive an epidural.
  Interventions: Other: Pulse oximeter
- Childbirth and general anesthesia: Pregnant women giving childbirth who receive general anesthesia
  Interventions: Other: Pulse oximeter
- Fetal Intervention and epidural: Pregnant women receiving fetal intervention and an epidural
  Interventions: Other: Pulse oximeter
- Fetal Intervention and general anesthesia: Pregnant women receiving fetal intervention and general anesthesia
  Interventions: Other: Pulse oximeter

INTERVENTIONS:
Other: Pulse oximeter — Place a pulse oximeter on the subject which will record the pulse oximeter waveform.

SUMMARY:
Using a pulse oximeter, the investigators have developed an algorithm that assesses central volume status. Pregnant women present some unique opportunities for us to investigate the algorithm under different circumstances. The investigators want to specifically investigate an algorithm with women who undergo regional anesthesia such as epidurals, with women who undergo fetal surgery, and with women in labor and giving birth (and the recovery time following delivery). This will help the investigators understand the central volume status changes that women experience in these unique circumstances. The Investigators also want to put the pulse oximeter on the fetal hand when possible during certain maternal fetal interventions. The Investigators would like to examine the algorithm with data from the fetuses.

DETAILED DESCRIPTION:
The Investigators hypothesize that the Compensatory Reserve Index (CRI) algorithm will help to guide fluid management in women undergoing regional anesthesia, giving birth, and/or undergoing maternal fetal intervention surgery.

Specific aims:

Collect noninvasive physiological waveform data from patients undergoing regional anesthesia and either fetal intervention surgery or labor and delivery at Children's Hospital Colorado in order to:

1. Determine how regional anesthesia influences CRI algorithm calculations
2. Determine if the CRI algorithm is able to detect changes in central volume status associated with fetal surgery.
3. Determine if the CRI algorithm is able to detect changes in central volume status associated with labor and childbirth specifically at the time of delivery, when most women experience some amount of bleeding.
4. Examine CRI associated with induction of regional anesthesia and determine if there is a minimal CRI below which one can expect hypotension and if there is a trend down in CRI following induction of regional anesthesia that could anticipate/predict hypotension.
5. Determine if there is a correlation between fetal heart rate abnormalities and CRI.
6. Examine CRI associated with fetal monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 14 years - 44 years or 0 day old neonates born during the protocol
2. Pregnant
3. Patients undergoing regional anesthesia and either fetal intervention surgery or labor at Children's Hospital Colorado (CHCO) or University of Colorado Hospital (UCH)

Exclusion Criteria:

1. Incarcerated
2. Decisionally challenged
3. Patients who object at any time to participating in the study

Ages: 0 Days to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Enrollment is limited to pregnant females because only pregnant females undergo fetal surgery and/or labor and childbirth.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-02-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Changes in Central Volume Status | enrollment
  Use pulse oximeter waveform data to determine central volume status changes

CONTACTS AND LOCATIONS:
Overall Officials: Steven Moulton, MD, Principal Investigator — Childrens Hospital Colorado